CLINICAL TRIAL: NCT04161963
Title: Incidence of Sub-clinical Cystoid Macular Edema After Cataract Surgery
Acronym: ICCME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ICCME
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cataract; Glaucoma
Keywords: Cataract; Glaucoma; cystroid macular edema
MeSH Terms: conditions — Cataract; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phaco: tandard ultrasound phacoemulsification cataract surgery
  Interventions: Device: SD-OCT; Device: OCT-A
- FLACS: femtolaser assisted cataract surgery
  Interventions: Device: SD-OCT; Device: OCT-A
- phaco+MIGS: combined phacoemulsification cataract surgery plus micro invasive glaucoma surgery
  Interventions: Device: SD-OCT; Device: OCT-A

INTERVENTIONS:
Device: SD-OCT — Optical Coherence Tomography of the maculy with Heidelberg Spectralis SD-OCT
Device: OCT-A — swept source Optical Coherence Tomography Angiography with Zeiss Plex Elite 9000 of the macula

SUMMARY:
Cystoid macular edema (CME) can limit visual acuity after cataract surgery. Little is known whether the incidence is similar between standard ultrasound phacoemulsification cataract surgery (phaco), femtolaser assisted cataract surgery (FLACS), and combined phacoemulsification cataract surgery plus micro invasive glaucoma surgery (phaco+MIGS) procedures.

DETAILED DESCRIPTION:
Subclinical cystoid macular edema (CME) can limit visual acuity after cataract surgery. Little is known whether the incidence is similar between standard ultrasound phacoemulsification cataract surgery (phaco), femtolaser assisted cataract surgery (FLACS), and combined phacoemulsification cataract surgery plus micro invasive glaucoma surgery (phaco+MIGS) procedures.

The investigators hypothesize that CME incidence will be in the following order: FLACS < phaco < phaco+MIGS due to the increase of inflammation with the different surgical procedures.

The study is designed as a single centre, prospective study. The study includes patients with a diagnosis of cataract or cataract and glaucoma who will undergo one of the three above mentioned sürgical procedures at the Department of Ophthalmology at the UniversityHospital Zurich (USZ), Zurich, Switzerland. CME will be assessed by optical coherence tomography of the macular with Heidelberg Spectralis SD-OCT of the Macular at: baseline (i.e. preoperative), 1 week, 1 month, 3 months, and 6 months post-surgery. Furthermore, a swept source Optical Coherence Tomography Angiography (OCT-A) using Zeiss Plex Elite 9000 will be performed at: baseline (i.e. preoperative), 1 week, 1 month, and 6 months post-surgery to image the retinal vessels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cataract or
* Patients with a diagnosis of cataract and open angle glaucoma
* Signed lnformed Consent
* Patients at the age of 18 or older

Exclusion Criteria:

* Loss of follow up, i.e. not available during the post-operation follow-up inteval.
* Previous known of CME, macular pathology (e.g., Diabetes, exudative age-related macular degeneration, status post retinal vein occlusion) or posterior uveitis.
* Patient unable to understand the study due to cognitive or linguistic incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who will undergo cataract surgery or combined catarct MIGS glaucoma surgery at the University Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of CME | baseline/preop
  incidence of subclinical cystoid macular edema
incidence of CME | 1 week postop +/- 4 days
  incidence of subclinical cystoid macular edema
incidence of CME | 1 month postop +/-2 weeks
  incidence of subclinical cystoid macular edema
incidence of CME | 3 months postop +/-2 weeks
  incidence of subclinical cystoid macular edema
incidence of CME | 6 months postop +/-2 weeks
  incidence of subclinical cystoid macular edema

CONTACTS AND LOCATIONS:
Overall Officials: Marc Töteberg-Harms, MD, FEBO, Principal Investigator — University Hospital Zurich, Department of Ophthalmology
Locations (1):
- Department of Ophthalmology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No